CLINICAL TRIAL: NCT02737345
Title: Correlation of Hepatitis C, Alcoholic Liver Disease, and Renal Failure With Hyperfibrinolysis in Liver Failure
Status: Completed | Type: Observational
Sponsor: Scott Allen (Other)
Responsible Party: Sponsor-Investigator, Scott Allen, Anesthesiologist, University of Utah
Organization: University of Utah (Other)
Other Study IDs: 00086371
Record Dates: First submitted 2016-04-01; First posted 2016-04-13 (Estimated); Last update posted 2017-11-08 (Actual); Status verified 2017-11

CONDITIONS: Cirrhosis
Keywords: fibrinolysis; liver transplant; thromboelastometry
MeSH Terms: conditions — Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Waiting list: Patients on the liver transplant waiting list
  Interventions: Other: Rotem

INTERVENTIONS:
Other: Rotem

SUMMARY:
1. Further characterize the incidence of hyperfibrinolysis in cirrhotics
2. Correlate hyperfibrinolysis with

   1. hepatitis C
   2. alcoholic liver disease
   3. the subset of a&b with renal failure with and without dialysis
3. Better describe the hyperfibrinolytic ROTEM profile in cirrhotics

ELIGIBILITY:
Inclusion Criteria:

* Be on the the liver transplant waiting list

Exclusion Criteria:

* liver failure without eligibility for transplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with liver failure who are on the liver transplant waiting list
Sampling Method: Non-Probability Sample
Enrollment: 54 (Actual)
Dates: Start 2015-11-01 (Actual); Primary Completion 2017-04-01 (Actual); Study Completion 2017-04-01 (Actual)

PRIMARY OUTCOMES:
The percentage of patients who exhibit fibrinolysis | Within 60 minutes of sample run time
  The percentage of patients who exhibit fibrinolysis, defined as a decrease in maximum clot firmness <15% within 60 minutes of sample run time.

CONTACTS AND LOCATIONS:
Overall Officials: Scott Allen, MD, Principal Investigator — University of Utah
Locations (1):
- University of Utah, Salt Lake City, Utah, United States